CLINICAL TRIAL: NCT03279692
Title: Phase II Trial of Pembrolizumab in Recurrent or Residual High Grade Meningioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Priscilla Brastianos, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-296
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: High Grade Meningioma
Keywords: Meningioma
MeSH Terms: conditions — Meningioma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): * Pembrolizumab will be administered every 3 weeks
  * Pembrolizumab will be administered through IV infusion
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab binds to PD-1, an inhibitory signaling receptor expressed on the surface of activated T cells, and blocks the binding to and activation of PD-1 by its ligands, which results in the activation of T-cell-mediated immune responses against tumor cells
  Other Names: Keytruda

SUMMARY:
This research study is studying a drug as a possible treatment for High Grade Meningioma.

The drug involved in this study is an immunotherapy drug called pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for this specific disease but it has been approved for other uses.

In this research study, the investigators are studying pembrolizumab in participants with meningioma. Research studies have shown that meningioma tumor cells express a gene called PD-L1. The investigators will be looking to determine whether the study drug may may stop meningioma tumors from growing.

ELIGIBILITY:
Inclusion Criteria:

-Documentation Of Disease

--Histologic Documentation: Histologically proven recurrent or residual intracranial or metastatic meningioma or meningioma with extracranial spread

Progressive OR residual disease, as defined by the following:

* Progressive disease, as defined as an increase in size of the measurable primary lesion on imaging by 25% or more (bidirectional area). The change must occur between scans separated by no more than 24 months.
* Residual measurable disease: For Grade II or III meningioma, residual measurable disease immediately after surgery without requirement for progression. Residual measurable disease will be defined by bidimensionally measurable lesions with clearly defined margins by MRI scans, with a minimum diameter of 10mm in both dimensions.
* Post radiation patients: Patients with measurable and progressive meningioma who have received radiation are potentially eligible, but need to show evidence of progressive disease in the radiated field after completion of radiation. At least 24 weeks must have elapsed from completion of radiation to registration. Patients that have progressive disease outside of the radiation field do not need to wait 24 weeks from completion of radiation.

  * Measurable Disease: Measurable disease is defined by a bidimensionally measurable main lesion on MRI or CT images (MRI preferred) with clearly defined margins and ≥ 10 mm. Multifocal disease is allowed as long as one lesion meets criteria for measurable disease and progressive disease.

Prior Treatment

* Prior medical therapy is allowed but not required.
* Meningioma that have resulted from prior radiation therapy are allowed.
* No limit on number of prior therapies.
* No chemotherapy, other investigational agents within 14 days of study treatment.
* No other concurrent investigational agents or other meningioma-directed therapy (chemotherapy, radiation) while on study.
* For patients treated with external beam radiation, interstitial brachytherapy or radiosurgery, an interval > 24 weeks must have elapsed from completion of XRT to registration.
* Stable dose of dexamethasone 2mg or less for 7 days prior to initiation of treatment
* Recovered to CTCAE grade 1 or less toxicity from other agents with exception of alopecia and fatigue.
* No craniotomy within 28 days of registration.

  * Not pregnant and not nursing:
  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months). Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
  * Age ≥ 18 years
  * ECOG Performance Status < 2
  * Patient history: Patients with history of NF may have other stable CNS tumors (schwannoma, acoustic neuroma or ependymoma) if lesions have been stable for 6 months.
  * Metastatic meningiomas (as defined by extracranial meningiomas) and meningioma with extra-cranial spread are allowed.
  * Required Initial Laboratory Values
  * Participants must have normal organ and marrow function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.
  * Required Initial Laboratory Values
* System Laboratory Value
* Hematological
* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL
* Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)

  -Renal
* Serum creatinine OR
* Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

  ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
* Albumin >2.5 mg/dL
* Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT)
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

  ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Creatinine clearance should be calculated per institutional standard.

  * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
  * Ability to understand and the willingness to sign a written informed consent document.
  * Stable dose of dexamethasone 2mg or less for 7 days prior to initiation of treatment

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days of protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Participants with brainstem lesions
* Participants who are receiving any other investigational agents.
* Participants who have a diagnosis of an immunodeficiency.
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone >2mg/day or bioequivalent within 7 days of initiating therapy.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids as described in Section 5.7, within three months of start of study drug
* Hypersensitivity to pembrolizumab or any of its excipients
* Has a known history of active TB (Bacillus Tuberculosis)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or stable NF-related neoplasms (Section 3.1.7).
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Unable to undergo brain MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Brastianos, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brastianos PK, Kim AE, Giobbie-Hurder A, Lee EQ, Wang N, Eichler AF, Chukwueke U, Forst DA, Arrillaga-Romany IC, Dietrich J, Corbin Z, Moliterno J, Baehring J, White M, Lou KW, Larson J, de Sauvage MA, Evancic K, Mora J, Nayyar N, Loeffler J, Oh K, Shih HA, Curry WT, Cahill DP, Barker FG, Gerstner ER, Santagata S. Phase 2 study of pembrolizumab in patients with recurrent and residual high-grade meningiomas. Nat Commun. 2022 Mar 14;13(1):1325. doi: 10.1038/s41467-022-29052-7. PMID 35289329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient withdrew consent before receiving pembrolizumab and was excluded from efficacy and safety analyses.
Groups:
- Pembrolizumab: * Pembrolizumab will be administered every 3 weeks
  * Pembrolizumab will be administered through IV infusion
  Pembrolizumab: pembrolizumab binds to PD-1, an inhibitory signaling receptor expressed on the surface of activated T cells, and blocks the binding to and activation of PD-1 by its ligands, which results in the activation of T-cell-mediated immune responses against tumor cells
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 26
Completed | 25
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months (PFS6)
Description: Progression-free survival at 6 months is defined as not having disease progression per RANO (response assessment in neuro-oncology) criteria or death from any cause within six months of the first day of treatment with pembrolizumab.
  Contrast-enhanced cranial magnetic resonance imaging (MRI) was performed every 6 weeks to assess patient response to treatment. Progressive disease is defined per RANO criteria as the appearance of a new lesion, an increase in the size of a patient's existing lesions, or clear clinical worsening (seizures, medication side effects, complications of therapy, cerebrovascular events, infection, etc.)
Time Frame: up to 6 months
Measure: Number (90% Confidence Interval); unit: percent of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
percent of participants | 48 [31 to 66]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from protocol registration until death due to any cause. The follow-up of patients who were alive at the time of analysis was censored at the date of last assessment of vital status. 90% confidence intervals for median OS were estimated using log(-log(survival)) methodology.
Time Frame: Up to 35 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
months | 20.2 [14.8 to 25.8]

3. Secondary Outcome: Overall Survival (OS) at 3 Months
Description: OS benchmarked at 3 months measures the percentage of participants who are still alive at 3 months, after study registration and receiving study therapy.
Time Frame: 3 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
percentage of participants | 92 [77 to 97]

4. Secondary Outcome: Overall Survival (OS) at 6 Months
Description: OS benchmarked at 6 months measures the percentage of participants who are still alive at 6 months, after study registration and receiving study therapy.
Time Frame: 6 months
Measure: Number (90% Confidence Interval); unit: percent of patients
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
percent of patients | 84 [67 to 93]

5. Secondary Outcome: Percentage of Participants With Treatment-related Adverse Events
Description: All adverse events (AEs) recorded during the trial were summarized for all patients who received one or more doses of pembrolizumab. This outcome measure includes adverse events assessed as at least possibly related to study therapy and grade 3 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: Up to 26 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
Participants | 20

6. Secondary Outcome: Number of Participants With Intracranial Response
Description: Intracranial response is defined as complete response (CR), partial response (PR), or stable disease (SD) by RANO (response assessment for neuro-oncology) criteria. Intracranial response was assessed by contrast-enhanced cranial magnetic resonance imaging (MRI) every 6 weeks.
  CR: complete disappearance of all enhancing measurable and non-measurable disease sustained for 4+ weeks, no new lesions, stable/decreasing corticosteroids, and patient is stable and improved clinically. Participants with non-measurable disease cannot have a CR; the best possible response is SD.
  PR: greater than or equal to 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for 4+ weeks, no progression of non-measurable disease, no new lesions, stable/decreasing corticosteroids, and patient is stable or improved clinically.
  SD: does not qualify for CR, PR, or disease progression and patient is stable clinically.
Time Frame: Up to 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 18

ADVERSE EVENTS:
Time Frame: up to 3 years
Description: In addition to the clinicaltrials.gov seriousness criteria, the following seriousness criteria are added: (1) new cancer (that is not a condition of the study) and (2) associated with an overdose.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 15/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=25)
Skin/subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Basal Cell Carcinoma
Seizure (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Generalized Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) — Cellulitis
Encephalopathy (Nervous system disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — Bifrontal Craniotomy
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Chronic Obstructive Pulmonary Disease Exacerbation
Anemia (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate Aminotransferase increased (Investigations) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Gallstone
Lung Infection (Infections and infestations) | 1 (1) — Pneumonia
Dysarthria (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=25)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 4 (4)
Alopecia (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — Intermittent Decreased Red Blood Cell Count
Blood bilirubin increased (Investigations) | 1 (1)
Blood corticotrophin decreased (Investigations) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — Systolic Murmur
Chills (General disorders) | 2 (2)
Cholesterol High (Investigations) | 7 (7)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Concentration Impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine Increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 2 (3)
Edema cerebral (Nervous system disorders) | 1 (1)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 5 (5)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (5) — eGFR abnormality
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — bandemia
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — Left Ventricular Outflow Tract Obstruction
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Neurotropic ulcer left eye
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Eye Discharge
Eye pain (Eye disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (18)
Fatigue (General disorders) | 12 (15)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 7 (9)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Diverticulosis
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Mouth Pain
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Thrush
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Ingrown toenail
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Postural Difficulty
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Left Arm Orbiting
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Left Pronator Drift
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Left Pointer Finger inflammation with Drainage
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Hypopituitarism
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Collapsed right nostril
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Upper Right Eyelid Lymphedema
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Right Brow Ptosis
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Right forearm lesion
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (7)
Headache (Nervous system disorders) | 4 (6)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — jaundice
Hyperglycemia (Metabolism and nutrition disorders) | 7 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (6)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (4)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Bilateral toe fungus
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Herpes simplex virus vesicle
Insomnia (Psychiatric disorders) | 7 (7)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (1) — Decreased free T4
Investigations - Other, specify (Investigations) | 1 (1) — Decreased free T3
Investigations - Other, specify (Infections and infestations) | 7 (8) — Elevated LDH
Investigations - Other, specify (Investigations) | 2 (2) — Elevated Neutrophil Count
Investigations - Other, specify (Investigations) | 1 (1) — TSH elevated
Investigations - Other, specify (Investigations) | 1 (1) — Free T4 Elevated
Lethargy (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5)
Lipase increased (Investigations) | 1 (1)
Localized edema (General disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5)
Memory impairment (Nervous system disorders) | 2 (2)
Investigations - Other, specify (Investigations) | 2 (2) — Decreased TSH
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Cramping, left leg
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Right ankle pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Right calf swelling
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Neck edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Adrenal Adenoma
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Numbness, face
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Hypertonicity (worsening)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Aura
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Staring Spells
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Facial twitch
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Left Ptosis
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Myoclonus
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Right Hemiparesis
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Dysmetria
Neutrophil count decreased (Investigations) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) — Panic Attack
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 4 (6)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) — Vaginal lesion
Upper Respiratory Infection (Infections and infestations) | 2 (2)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 6 (10)
Serum amylase increased (Investigations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Nail irritation
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Scalp swelling
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Atypical squamous proliferation
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Benign Seborrheic Keratoses
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Actinic keratoses
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Verruca vulgaris
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Scaly skin irritation
Truncal rash (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spasticity (Nervous system disorders) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Urinary Incontinence (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) — Atheroma
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03279692/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03279692/ICF_001.pdf